CLINICAL TRIAL: NCT00353574
Title: DORADO-EX - A Dose-Blinded, Long-Term Safety Extension Study of Fixed Doses of Darusentan in Subjects With Resistant Systolic Hypertension Receiving Combination Therapy With Three or More Antihypertensive Drugs, Including a Diuretic (Protocol DAR-311-E)
Brief Title: DORADO-EX: Long-Term Safety Extension Study to the Phase 3 DORADO Study (Protocol DAR-311) of Darusentan in Resistant Hypertension
Acronym: Darusentan
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study DAR-312 did not meet primary co-endpoints
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DAR-311-E
Record Dates: First submitted 2006-07-17; First posted 2006-07-18 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-02

CONDITIONS: Hypertension
Keywords: Resistant Hypertension
MeSH Terms: conditions — Hypertension | interventions — darusentan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Darusentan 50 mg (Experimental): Darusentan 50 mg administered orally once daily
  Interventions: Drug: Darusentan
- Darusentan 100 mg (Experimental): Darusentan 100 mg administered orally once daily
  Interventions: Drug: Darusentan
- Darusentan 300 mg (Experimental): Darusentan 300 mg administered orally once daily
  Interventions: Drug: Darusentan

INTERVENTIONS:
Drug: Darusentan — Darusentan capsules administered orally once daily

SUMMARY:
This is a research study of a new experimental drug called darusentan. Darusentan is not currently approved by the United States (U.S.) Food and Drug Administration (FDA) for use in the U.S., which means that a doctor cannot prescribe this drug. The purpose of this study is to evaluate the long-term safety of darusentan in subjects with resistant systolic hypertension despite treatment with full doses of three or more antihypertensive medications, including a diuretic.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have completed the Treatment Period of clinical trial DAR-311
* Receiving and adhering to full doses of appropriate guideline-recommended antihypertensive drugs from three different classes of antihypertensive agents, including a diuretic

Exclusion Criteria:

* Subjects who discontinued treatment with study drug prior to the end of the Treatment Period of DAR-311 due to a study drug-related adverse event (AE)
* Treatment with another endothelin receptor antagonist within 6 months of study entry

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2006-09; Primary Completion 2010-02 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Change in trough sitting systolic and diastolic blood pressure | Baseline to Week 14

SECONDARY OUTCOMES:
Change in mean 24-hour systolic and diastolic ambulatory blood pressures. | Baseline to Week 14
Percentage of subjects who reach systolic blood pressure goal | Week 14
Change in estimated glomerular filtration rate (eGFR) | Baseline to Week 14

CONTACTS AND LOCATIONS:
Locations (75):
- United States (53):
  - Comprehensive Heart Failure Center, Mobile, Alabama
  - Canyon Clinical Research, Tucson, Arizona
  - Chrishard Medical Group, Inglewood, California
  - VA Medical Center - WLA, Los Angeles, California
  - Sacramento Heart and Vascular, Sacramento, California
  - Apex Research Institute, Santa Ana, California
  - Complete Renal Care, Denver, Colorado
  - Connecticut Clinical Research, LLC, Bridgeport, Connecticut
  - MedStar Diabetes Institute at Washington Hospital Center, Washington D.C., District of Columbia
  - White-Wilson Medical Center, Fort Walton Beach, Florida
  - A.G.A. Clinical Trials, Hialeah, Florida
  - Jacksonville Center for Clinical, Jacksonville, Florida
  - Ricardo A. Bedoya, Cardiology, Jupiter, Florida
  - International Research Association, Miami, Florida
  - Cardiovascular Center of Sarasota, Sarasota, Florida
  - Tampa Bay Nephrology Associates, PL, Tampa, Florida
  - Metabolic Research Institute, Inc., West Palm Beach, Florida
  - Global Research Partners, Calhoun, Georgia
  - Kula Research, Honolulu, Hawaii
  - Chicago Heart & Vein Clinic, Elk Grove Village, Illinois
  - Evanston Northwestern Healthcare, Evanston, Illinois
  - Clinical Investigation Specialists, Inc., Gurnee, Illinois
  - Midwest Heart Foundation, Lombard, Illinois
  - Medical Research Institute, Slidell, Louisiana
  - Androscoggin Cardiology Associates, Auburn, Maine
  - Maine Research Associate, Auburn, Maine
  - Cardiovascular Consultants of Maine, Scarborough, Maine
  - Clinical Associates, Reisterstown, Maryland
  - Rockville Internal Medicine Group, Rockville, Maryland
  - Professional Clinical Research, Benzonia, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Professional Clinical Research, Interlochen, Michigan
  - Specialty Medical Center, Pahrump, Nevada
  - Physicians East, PA, Greenville, North Carolina
  - The Lindner Clinical Trial Center, Cincinnati, Ohio
  - COR Clinical Research, Oklahoma City, Oklahoma
  - Southwest Cardiology Associates, Oklahoma City, Oklahoma
  - Castlerock Clinical Research Consultants, Tulsa, Oklahoma
  - Hillsboro Cardiology, PC, Hillsboro, Oregon
  - Northeast Clinical Research Centers, Inc., Allentown, Pennsylvania
  - Heritage Cardiology Associates, Camp Hill, Pennsylvania
  - Brandywine Clinical Research, Downingtown, Pennsylvania
  - Green and Seidner Family Practice Associates, Lansdale, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - RI Hospital, Providence, Rhode Island
  - Neem Research Group, Inc., Columbia, South Carolina
  - Internal Medicine & Industrial Medicine, DeSoto, Texas
  - T&R Clinical, P.A., Fort Worth, Texas
  - Pri-Med Care, Lewisville, Texas
  - Innovative Clinical Trials, San Antonio, Texas
  - Burke Internal Medicine, Inc., Burke, Virginia
  - Manassas Clinical Research Center, Manassas, Virginia
  - Liberty Research Center, Tacoma, Washington
- Argentina (8):
  - CIMEL, Buenos Aires
  - DIM (Clinica Privada), Buenos Aires
  - Fundapres, Buenos Aires
  - Hospital Britanico de Buenos Aires, Buenos Aires
  - Hospital Jose Maria Ramos Meijia, Buenos Aires
  - Hospital Municipal Bernardo Houssay, Buenos Aires
  - Medeos, Buenos Aires
  - Sanatorio Municipal, Buenos Aires
- Brazil (2):
  - Centro Integrado Hospital do Rim e Hipertensao, São Paulo
  - Centro Integrado Hospital, São Paulo
- Canada (2):
  - Cambridge Cardiac Care Center, Cambridge, Ontario
  - Clinical Research Solutions, Kitchener, Ontario
- Denmark (2):
  - Bispebjerg Hospital, Copenhagen
  - Hvidovre Hospital, Hvidovre
- France (3):
  - CIC Hopital Jeanne D'Arc, Dommartin-lès-Toul
  - CHU de Grenoble, Grenoble
  - Hôpital Civil, Service HTA maladies vasculaires, Strasbourg
- Sweden (2):
  - Cardiovascular Research, Karolinska Institue, Stockholm
  - University Hospital Umea, Umeå
- United Kingdom (3):
  - Townhead Surgery, Scotland
  - Avenue Surgery, Wiltshire
  - Hathaway Medical Centre, Wiltshire

REFERENCES:
- See also: Related Info — http://www.gilead.com